CLINICAL TRIAL: NCT03837717
Title: The Impact of Holding During Therapeutic Hypothermia on Saliva Oxytocin and Cortisol Levels in Mother-Infant Pairs
Brief Title: The Impact of Holding on Stress and Bonding in Mother-Infant Pairs During Therapeutic Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Alexa Craig, Attending Pediatric Neurologist, MaineHealth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1183063
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2019-10

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Neonatal Encephalopathy
Keywords: Saliva; Neonatal Encephalopathy; Hypoxic-Ischemic Encephalopathy; Bonding; Oxytocin; Stress; Cortisol
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: Infants and mothers will be randomly assigned to the holding condition occurring on the second versus the third day of hypothermia.
  On the day of holding, four samples of saliva will be obtained; two from the mother (pre and post holding) and two from the infant (pre and post holding). The first sample will be collected prior to holding, and the second sample immediately at the end of holding before the infant is placed back in the bed.
  On the day without holding, four additional samples of saliva will be obtained; two from the mother (pre and post "not holding") and two from the infant (pre and post "not holding").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holding First (Experimental): Holding will occur on the second day of hypothermia treatment. Saliva will be collected on Day 2 and Day 3
  Interventions: Behavioral: Holding; Other: Saliva collection; Behavioral: No Holding
- No Holding First (Experimental): Holding will occur on the third day of hypothermia treatment. Saliva will be collected on Day 2 and Day 3
  Interventions: Behavioral: Holding; Other: Saliva collection; Behavioral: No Holding

INTERVENTIONS:
Behavioral: Holding — Mothers will be assisted with holding their infants (and the cooling blanket) for a single 30-minute period, with the use of a thin foam barrier for thermal protection. Mothers and infants will not be skin-to-skin.
Other: Saliva collection — Saliva will be collected from infants (via syringe suction) and mothers (via passive drool), and tested for levels of cortisol and oxytocin
Behavioral: No Holding — Saliva will be collected from Mothers and infants, and vital sign information will be collected from infants in the same manner as the Holding intervention, with the exception of having mother's hold their infants.

SUMMARY:
This research is being done to try to improve the experience of mothers and babies during therapeutic hypothermia. Currently, mothers are not able to hold their baby during hypothermia treatment. Mothers have reported that not being able to hold their baby during this time is stressful. Additionally, it is known that holding has many benefits for mothers' and babies' psychological and physical health.

Therapeutic hypothermia is the standard of care. The experimental interventions of this study are to have mothers hold their babies during this treatment, collect saliva samples from mothers and babies, and test the saliva samples for the hormones cortisol and oxytocin. The investigators will test saliva of infants and their mothers before and after holding. The investigators hope to demonstrate decreased cortisol, a marker for stress, and increased oxytocin, a marker for bonding, in infants and mothers while they are held during therapeutic hypothermia.

DETAILED DESCRIPTION:
The inability to hold an infant being treated with therapeutic hypothermia in the neonatal intensive care unit has been subjectively reported by ours and other research groups as a significant source of stress for parents. The investigators aim to assess the impact of holding on endocrinological markers of stress and bonding. Specifically, the investigators plan to collect salivary cortisol and oxytocin levels from infants undergoing therapeutic hypothermia and their mothers prior to and immediately after a 30-minute holding period.

The investigators hypothesize that measurable increases in salivary oxytocin levels, coinciding with the reported qualitative increased levels of bonding, will be observed after the holding period. The investigators anticipate the reported stress reduction after holding to be quantified by measurable decreases in salivary cortisol levels. The investigators hypothesize these hormone changes will be present in both the mother and the infant when compared to samples taken without the holding intervention.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth of 35 weeks or greater
* absence of clinical or electrographic seizures during the first 24 hours of therapeutic hypothermia
* designation as "clinically stable" by the attending neonatologist on service
* respiratory status of: room air, nasal cannula, continuous positive airway pressure or intubated on conventional ventilator

Exclusion Criteria:

* designation as "clinically unstable" by the a member of the medical team
* use of inhaled nitric oxide for persistent pulmonary hypertension of the newborn
* high frequency oscillator ventilation
* presence of electrographic seizures
* use of vasopressors or paralytic agents, presence of chest tubes, wound vacuums, or drains
* in utero opiate exposure

Ages: 24 Hours to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Change in the level of oxytocin in maternal saliva | 30-minutes
  To compare the change in the level of oxytocin in maternal saliva between two conditions; one assessing the difference between oxytocin levels before and immediately after a 30-minute period of holding during therapeutic hypothermia compared to the second condition in which pre and post-levels of salivary oxytocin surrounding a 30-minute period of "not holding" are obtained.

SECONDARY OUTCOMES:
Change in the level of cortisol in maternal saliva | 30-minutes
  To compare the change in the level of cortisol in maternal saliva between two conditions; one assessing the difference between cortisol levels before and immediately after a 30-minute period of holding during therapeutic hypothermia compared to the second condition in which pre and post-levels of salivary cortisol surrounding a 30-minute period of "not holding" are obtained.
Change in the level of oxytocin and cortisol in infant saliva | 30-minutes
  To compare the change in the level of oxytocin and cortisol in infant saliva between the same two conditions
Comparison of infant temperature before, during and after holding | 30 minutes prior to holding, 30 minutes during holding, and 45 minutes after holding.
  Comparison between the holding and "not holding" conditions of infant temperature in °C, collected 30 minutes prior to holding, every 2 minutes during, and 45 minutes after holding.
Comparison of infant heart rate before, during and after holding | 30 minutes prior to holding, 30 minutes during holding, and 45 minutes after holding.
  Comparison between the holding and "not holding" conditions of infant heart rate in beats per minute, collected 30 minutes prior to holding, every 2 minutes during, and 45 minutes after holding.
Comparison of infant blood pressure before, during and after holding | 30 minutes prior to holding, 30 minutes during holding, and 45 minutes after holding.
  Comparison between the holding and "not holding" conditions of infant mean arterial blood pressure, measured with an arterial line, or, if none present, with systolic and diastolic cuff pressures, collected 30 minutes prior to holding, every 2 minutes during, and 45 minutes after holding.
Comparison of infant oxygen saturation before, during and after holding | 30 minutes prior to holding, 30 minutes during holding, and 45 minutes after holding.
  Comparison between the holding and "not holding" conditions of infant percent oxygen saturation collected 30 minutes prior to holding, every 2 minutes during, and 45 minutes after holding.
Subjective maternal reports | Immediately after 30-minutes of holding
  Subjective maternal reports of the experience of holding the infant during hypothermia and responses to questions about stress level and bonding.
Subjective nurse reports | Immediately after 30-minutes of holding
  Subjective nurse report about the experience of assisting with holding.

CONTACTS AND LOCATIONS:
Overall Officials: Alexa K Craig, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vittner D, McGrath J, Robinson J, Lawhon G, Cusson R, Eisenfeld L, Walsh S, Young E, Cong X. Increase in Oxytocin From Skin-to-Skin Contact Enhances Development of Parent-Infant Relationship. Biol Res Nurs. 2018 Jan;20(1):54-62. doi: 10.1177/1099800417735633. Epub 2017 Oct 11. PMID 29017336
- [Background] Craig AK, James C, Bainter J, Evans S, Gerwin R. Parental perceptions of neonatal therapeutic hypothermia; emotional and healing experiences. J Matern Fetal Neonatal Med. 2020 Sep;33(17):2889-2896. doi: 10.1080/14767058.2018.1563592. Epub 2019 Jan 8. PMID 30585100
- [Background] Craig AK, Gerwin R, Bainter J, Evans S, James C. Exploring parent expectations of neonatal therapeutic hypothermia. J Perinatol. 2018 Jul;38(7):857-864. doi: 10.1038/s41372-018-0117-8. Epub 2018 May 8. PMID 29740186
- [Background] Craig AK, Gerwin R, Bainter J, Evans S, James C. Exploring Parent Experience of Communication About Therapeutic Hypothermia in the Neonatal Intensive Care Unit. Adv Neonatal Care. 2018 Apr;18(2):136-143. doi: 10.1097/ANC.0000000000000473. PMID 29595551
- [Background] Craig A, Deerwester K, Fox L, Jacobs J, Evans S. Maternal holding during therapeutic hypothermia for infants with neonatal encephalopathy is feasible. Acta Paediatr. 2019 Sep;108(9):1597-1602. doi: 10.1111/apa.14743. Epub 2019 Mar 5. PMID 30721531

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT03837717/Prot_SAP_000.pdf